CLINICAL TRIAL: NCT02161900
Title: Randomized Controlled Trial Evaluating the Role of Exercise in Women Undergoing Treatment for Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Rajendra A. Badwe, Director, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMH Project No. 735
Record Dates: First submitted 2014-05-20; First posted 2014-06-12 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Non Metastatic Operable Breast Cancer

STUDY DESIGN:
Intervention Model Description: Yogic exercises are being evaluated for better supportive care over standard exercises for the breast cancer patients under treatment
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine exercise (Active Comparator): All newly diagnosed cases with stage I-III of breast cancer who present to Tata Memorial Hospital will be randomly assigned to perform either a set of 'Yogic and Routine Exercises (referred to as exercise I) or Routine Exercises'(referred to as exercise II) . Patients will begin the exercises within a week of starting treatment.
  Interventions: Other: Yogic and routine exercises
- Yogic and Routine exrcises (exercise I) (Experimental): All newly diagnosed cases with stage I-III of breast cancer who present to Tata Memorial Hospital will be randomly assigned to perform either a set of 'Yogic and Routine Exercises (referred to as exercise I) or Routine Exercises'(referred to as exercise II) . Patients will begin the exercises within a week of starting treatment.
  Interventions: Other: Yogic and routine exercises

INTERVENTIONS:
Other: Yogic and routine exercises — All newly diagnosed cases with stage I-III of breast cancer who present to Tata Memorial Hospital will be randomly assigned to perform either a set of 'Yogic and Routine Exercises (referred to as exercise I) or Routine Exercises'(referred to as exercise II) . Patients will begin the exercises within a week of starting treatment.

SUMMARY:
TITLE: Randomized Controlled Evaluating the Role of Exercise in Women Undergoing Treatment for Breast Cancer

Yoga and Quality of life:

Yoga is based on the practice of physical postures, breathing techniques and meditation. Philosophically, it aims at increasing the body's ability to master the mind with the goal of spiritual awareness and connection. A randomized trial of yoga in women with breast cancer undergoing radiation therapy demonstrated an improvement in impact of events scale at 3 months suggesting that the more intrusive thoughts at 1 month the greater the finding of meaning in cancer by 3 months. Randomized studies have demonstrated evidence of yoga improving the emotional well being of women with breast cancer and improving their distressed mood, thus providing a buffering effect on QOL. The main beneficial effects demonstrated are on social functioning. Among patients not receiving chemotherapy, yoga appears to enhance emotional well-being and mood and may serve to buffer deterioration in both overall and specific domains of QOL.

EVALUATION TOOLS- European Organisation for Research and Treatment of Cancer-Quality of Life Questionnaire (EORTC QLQ-C30 & BR-23) Brief Fatigue Inventory VAS (Pain score) Spirituality Questionnaire Pulmonary function test Objective assessment

STUDY ENDPOINTS- Primary end points- Disease free survival Secondary end points- Quality of life & Improvements in overall survival

STUDY DESIGN TREATMENT PLAN - All newly diagnosed cases with stage I-III of breast cancer who present to Tata Memorial Hospital will be randomly assigned to perform either a set of 'Yogic and Routine Exercises (referred to as exercise I) or Routine Exercises'(referred to as exercise II)./ Patients will begin the exercises within a week of starting treatment.

Both arms of the study will receive a training session one hour per day for the first week, during which they will be instructed to practice daily and maintain a daily log. The other evaluation tools will be used as per the assessment time line (enclosed).The exercises in the Exercise I arm (Yoga and conventional exercises) will be upgraded within the next 2 days to Phase II. Patients will be allowed to attend a minimum of four out of seven days in Phase I and II. Patients will be assessed at 6 months for compliance to phase II exercises. Only if patients are fulfilling the criteria for accuracy, sequence and duration of phase II exercises, will they be taught phase III exercises. Patients who are unable to do phase II exercises at 6 months will be re taught phase II exercises. These patients will then be re assessed at 1 year for up gradation to phase III. Six months after completion of phase III exercises, patients will be assessed for compliance to phase III exercises. Patients will also undergo an objective assessment at 1 year. An additional up gradation will be after completion of adjuvant therapy at 6 months.

Patients will be followed up for a period of 5 years. DFS will be measured from the time of randomization to either progression or death. Quality of life will be measured at baseline and every six monthly using the functional assessment cancer therapy- quality of life. Quality of Life analysis at 400 patients will be performed with appropriate correction for multiple analyses applied.

STATISTICAL ANALYSIS- For an expected 50% 5 year disease free survival (DFS) for the control group, the expected 5 years DFS for the intervention group will be 60%. With a two-sided analysis, and at 80% power and 95% confidence to detect a 10% difference between the arms, the sample size would be 761 patients. Assuming a 10% loss to follow up, a total of 850 patients would be accrued. We expect to complete accrual in 3 year.

RANDOMIZATION AND STRATIFICATION- Randomization for intervention will be done centrally from Clinical Research Secretariat and patient will be stratified by

Menopausal status: Pre + Peri or Post Neoadjuvant or adjuvant treatment Stage of disease: I/II/III ANALYSIS- Disease Free Survival (DFS) will be calculated from the date of randomization to the date of local, regional or distant relapse or death from any cause and will be censored at the last date of follow up for the patients that are alive and disease free or have been lost to follow up.

Overall Survival (OS) will be calculated from the date of randomization to the date of death or censored at the date of last follow up for the patients who are alive or lost to follow up. DFS and OS will be evaluated using Kaplan Meier and compared by Log-rank test. The Cox proportional hazard model will be used to assess the impact of intervention after correction for stratification, menopausal status and age.

ELIGIBILITY:
Inclusion Criteria:

* Women with unilateral breast cancer
* Age 18-65 years

Exclusion Criteria:

* Metastatic breast cancer
* Pregnant Women
* Women with physical limitations to perform exercises
* Previous history of cancer

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2010-11-12 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 5 years

SECONDARY OUTCOMES:
Quality of life, Improvements in overall survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India